CLINICAL TRIAL: NCT04432103
Title: Treatment of Severe and Critical COVID-19 Pneumonia With Convalescent Plasma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There is new evidence that the Convalescent plasma is not useful for severe and critical COVID-19 Pneumonia
Sponsor: Centro Medico ABC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC-20-14
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Covid-19
Keywords: covid-19; pneumonia; pandemic; convalescent plasma
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Two groups depending on the stage of the disease according to the CDC of China classification severe and critical COVID-19 pneumonia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe COVID-19 pneumonia (Experimental): Hospitalized patients with SARS-CoV 2 severe infection will receive an anti SARS-CoV 2 Convalescent Plasma
  Interventions: Biological: Anti SARS-CoV 2 Convalescent Plasma in severe COVID-19 patients
- Critical COVID- 19 pneumonia (Experimental): Hospitalized patients with SARS-CoV 2 critical infection will receive an anti SARS-CoV 2 Convalescent Plasma
  Interventions: Biological: Anti SARS-CoV 2 Convalescent Plasma in critical COVID-19 patients

INTERVENTIONS:
Biological: Anti SARS-CoV 2 Convalescent Plasma in severe COVID-19 patients — Administration of Convalescent Plasma to COVID-19 obtained from donors with prior documented SARS-CoV 2 infection with IgG antibodies to hospitalized COVID-19 severe cases.
  Arms: Severe COVID-19 pneumonia
Biological: Anti SARS-CoV 2 Convalescent Plasma in critical COVID-19 patients — Administration of Convalescent Plasma to COVID-19 obtained from donors with prior documented SARS-CoV 2 infection with IgG antibodies to hospitalized COVID-19 critical cases.
  Arms: Critical COVID- 19 pneumonia

SUMMARY:
Open label two arms, non randomized Convalescent Plasma treatment to severe and critical pneumonia COVID-19 hospitlaized patients compared to a historical cohort with matched controls.

DETAILED DESCRIPTION:
We will perform an open label two arms, non randomized trial giving Convalescent Plasma donated from recovered COVID-19 patients with positive serology to severe and clinical pneumonia COVID-19 patients admitted to the ABC Medical Center.

ELIGIBILITY:
Inclusion Criteria:

Donors:

1. Age: >18 and <60 years
2. Body weight : >60 kg
3. Confirmed previous SARS CoV-2 infection
4. negative SARS CoV-2 test result
5. 21 day without symptoms from the negative SARS CoV2 negative test
6. Written informed consent to participate in this clinical trial, to donate plasma and to store the specimen for future testing.
7. Positive COVID-19 IgG antibodies
8. Male donors, or female donors who have not been pregnant, or female donors who have been pregnant tested negative for HLA antibodies
9. Individuals who meet all regular voluntary donor eligibility requirements by the Mexican legislation.

Patients/recipients:

1. Age: >18 years
2. Admitted to the ABC Medical Center facility for the treatment of COVID-19
3. Patients with severe or critical COVID-19
4. Informed consent provided by the patient or healthcare proxy

Exclusion Criteria:

Patients/recipients:

1. Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products) 2. Any other not controlled infection 3. Disseminated Intravascular Coagulopathy 4. Patient under dialysis 5. Patient with recent Hemorrhagic Stroke 6. Severe Ischemic Heart Disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
INCIDENCE OF CRITICAL PNEUMONIA | 14 days after convalescent plasma administration
  progression to critical stage
MORTALITY RATE AMONG CRITICAL PNEUMONIA PATIENTS | 28 days after convalescent plasma administration
  mortality

SECONDARY OUTCOMES:
INCIDENCE OF MECHANICAL VENTILATION | 14 days after convalescent plasma treatment
  time to need mechanical ventilation
DAYS OF MECHANICAL VENTILATION | 28 days after convalescent plasma treatment
  time of mechanical ventilation needed

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Moreno, MD, Principal Investigator — ABC Medical Center Internal Medicine Department. Mexico City, Mexico; Irma Hoyo, MD PHD, Principal Investigator — ABC Medical Center Internal Medicine Department. Mexico City, Mexico; Benjamín Valente, MD MSc DTMH, Principal Investigator — ABC Medical Center Internal Medicine Department. Mexico City, Mexico
Locations (1):
- Centro Medico Abc, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Result] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Result] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Result] Burke RM, Midgley CM, Dratch A, Fenstersheib M, Haupt T, Holshue M, Ghinai I, Jarashow MC, Lo J, McPherson TD, Rudman S, Scott S, Hall AJ, Fry AM, Rolfes MA. Active Monitoring of Persons Exposed to Patients with Confirmed COVID-19 - United States, January-February 2020. MMWR Morb Mortal Wkly Rep. 2020 Mar 6;69(9):245-246. doi: 10.15585/mmwr.mm6909e1. PMID 32134909
- [Result] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643
- [Result] Rothe C, Schunk M, Sothmann P, Bretzel G, Froeschl G, Wallrauch C, Zimmer T, Thiel V, Janke C, Guggemos W, Seilmaier M, Drosten C, Vollmar P, Zwirglmaier K, Zange S, Wolfel R, Hoelscher M. Transmission of 2019-nCoV Infection from an Asymptomatic Contact in Germany. N Engl J Med. 2020 Mar 5;382(10):970-971. doi: 10.1056/NEJMc2001468. Epub 2020 Jan 30. No abstract available. PMID 32003551
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Result] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Liu K, Fang YY, Deng Y, Liu W, Wang MF, Ma JP, Xiao W, Wang YN, Zhong MH, Li CH, Li GC, Liu HG. Clinical characteristics of novel coronavirus cases in tertiary hospitals in Hubei Province. Chin Med J (Engl). 2020 May 5;133(9):1025-1031. doi: 10.1097/CM9.0000000000000744. PMID 32044814
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Patel A, Jernigan DB; 2019-nCoV CDC Response Team. Initial Public Health Response and Interim Clinical Guidance for the 2019 Novel Coronavirus Outbreak - United States, December 31, 2019-February 4, 2020. MMWR Morb Mortal Wkly Rep. 2020 Feb 7;69(5):140-146. doi: 10.15585/mmwr.mm6905e1. PMID 32027631
- [Result] Lu H. Drug treatment options for the 2019-new coronavirus (2019-nCoV). Biosci Trends. 2020 Mar 16;14(1):69-71. doi: 10.5582/bst.2020.01020. Epub 2020 Jan 28. PMID 31996494
- [Result] Kraft CS, Hewlett AL, Koepsell S, Winkler AM, Kratochvil CJ, Larson L, Varkey JB, Mehta AK, Lyon GM 3rd, Friedman-Moraco RJ, Marconi VC, Hill CE, Sullivan JN, Johnson DW, Lisco SJ, Mulligan MJ, Uyeki TM, McElroy AK, Sealy T, Campbell S, Spiropoulou C, Stroher U, Crozier I, Sacra R, Connor MJ Jr, Sueblinvong V, Franch HA, Smith PW, Ribner BS; Nebraska Biocontainment Unit and the Emory Serious Communicable Diseases Unit. The Use of TKM-100802 and Convalescent Plasma in 2 Patients With Ebola Virus Disease in the United States. Clin Infect Dis. 2015 Aug 15;61(4):496-502. doi: 10.1093/cid/civ334. Epub 2015 Apr 22. PMID 25904375
- [Result] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Result] Florescu DF, Kalil AC, Hewlett AL, Schuh AJ, Stroher U, Uyeki TM, Smith PW. Administration of Brincidofovir and Convalescent Plasma in a Patient With Ebola Virus Disease. Clin Infect Dis. 2015 Sep 15;61(6):969-73. doi: 10.1093/cid/civ395. Epub 2015 May 19. PMID 25991468
- [Result] Zhou B, Zhong N, Guan Y. Treatment with convalescent plasma for influenza A (H5N1) infection. N Engl J Med. 2007 Oct 4;357(14):1450-1. doi: 10.1056/NEJMc070359. No abstract available. PMID 17914053
- [Result] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Result] Burnouf T, Radosevich M. Treatment of severe acute respiratory syndrome with convalescent plasma. Hong Kong Med J. 2003 Aug;9(4):309; author reply 310. No abstract available. PMID 12904626
- [Result] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Result] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Result] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Result] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Result] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945
- [Result] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Result] Bloch EM, Shoham S, Casadevall A, Sachais BS, Shaz B, Winters JL, van Buskirk C, Grossman BJ, Joyner M, Henderson JP, Pekosz A, Lau B, Wesolowski A, Katz L, Shan H, Auwaerter PG, Thomas D, Sullivan DJ, Paneth N, Gehrie E, Spitalnik S, Hod EA, Pollack L, Nicholson WT, Pirofski LA, Bailey JA, Tobian AA. Deployment of convalescent plasma for the prevention and treatment of COVID-19. J Clin Invest. 2020 Jun 1;130(6):2757-2765. doi: 10.1172/JCI138745. PMID 32254064
- [Result] O'Shaughnessy DF, Atterbury C, Bolton Maggs P, Murphy M, Thomas D, Yates S, Williamson LM; British Committee for Standards in Haematology, Blood Transfusion Task Force. Guidelines for the use of fresh-frozen plasma, cryoprecipitate and cryosupernatant. Br J Haematol. 2004 Jul;126(1):11-28. doi: 10.1111/j.1365-2141.2004.04972.x. PMID 15198728
- See also: WHO Director-General's remarks at the media briefing on 2019-nCoV on 11 February 2020 [Internet]. [cited 2020 Mar 23]. — https://www-who-int.sire.ub.edu/dg/speeches/detail/who-director-general-s-remarks-at-the-media-briefing-on-2019-ncov-on-11-february-2020
- See also: Johns Hopkins Coronavirus Resource Center [Internet]. Johns Hopkins Coronavirus Resource Center. [cited 2020 Mar 23]. — http://coronavirus.jhu.edu/
- See also: Situation update worldwide, as of 22 March 2020 [Internet]. European Centre for Disease Prevention and Control. [cited 2020 Mar 23] — http://www.ecdc.europa.eu/en/geographical-distribution-2019-ncov-cases
- See also: Novel Coronavirus (2019-nCoV) situation reports [Internet]. [cited 2020 Mar 23]. — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports
- See also: who-china-joint-mission-on-covid-19-final-report.pdf [Internet]. [cited 2020 Mar 23]. — http://www-who-int.sire.ub.edu/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf
- See also: CDC. Coronavirus Disease 2019 (COVID-19) [Internet]. Centers for Disease Control and Prevention. 2020 [cited 2020 Apr 7]. — http://www-cdc-gov.sire.ub.edu/coronavirus/2019-ncov/hcp/clinical-criteria.html
- See also: National COVID-19 Convalescent Plasma Project [Internet]. [cited 2020 Apr 8]. — https://ccpp19.org/
- See also: Convalescent Plasma COVID-19 (Coronavirus) Treatment - Mayo Clinic [Internet]. [cited 2020 Apr 8]. Available from: — https://www.uscovidplasma.org/